CLINICAL TRIAL: NCT00977769
Title: Hemodynamic Effects of Carbetocin 100 µg, Oxytocin 5 U or Placebo After Cesarean Delivery Under Spinal Anesthesia in Healthy Pregnant Women.
Brief Title: Carbetocin Versus Oxytocin and Hemodynamic Effects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Leiv Arne Rosseland, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009carb
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-04

CONDITIONS: Effects of; Anesthesia, in Pregnancy
Keywords: cesarean delivery; blood pressure; cardiac output
MeSH Terms: interventions — carbetocin; Injections; Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- carbetocin 100 µg (Experimental): Carbetocin injection, 100µg, single injection
  Interventions: Drug: carbetocin 100 µg
- oxytocin 5 u (Active Comparator): Oxytocin 5U, injection, single injection
  Interventions: Drug: oxytocin 5 u
- placebo (NaCl) (Placebo Comparator): Saline single injection
  Interventions: Drug: placebo (NaCl)

INTERVENTIONS:
Drug: carbetocin 100 µg — Hemodynamic effect of
  Other Names: Pabal, injection
  Arms: carbetocin 100 µg
Drug: oxytocin 5 u — Hemodynamic effect of
  Other Names: Syntocinon, injection
  Arms: oxytocin 5 u
Drug: placebo (NaCl) — Hemodynamic effect of
  Other Names: Saline, injection
  Arms: placebo (NaCl)

SUMMARY:
A randomized double-blind trial of oxytocin 5 u, carbetocin 100 µg and placebo with hemodynamic response as a primary outcome measure.

DETAILED DESCRIPTION:
Healthy pregnant women sheduled for elective cesarean section. Invasive hemodynmaic monitoring with LiDCO Plus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women for planned cesarean section

Exclusion Criteria:

* Bleeding disorders
* Placenta disorders

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leiv Arne Rosseland, MD PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Division of Anaesthesia and Intensive Care Medicine, Oslo University Hospital - Rikshospitalet, Oslo
  - Division of Anesthesia and Intensive Care Medicine, Oslo

REFERENCES:
- [Result] Rosseland LA, Hauge TH, Grindheim G, Stubhaug A, Langesaeter E. Changes in blood pressure and cardiac output during cesarean delivery: the effects of oxytocin and carbetocin compared with placebo. Anesthesiology. 2013 Sep;119(3):541-51. doi: 10.1097/ALN.0b013e31829416dd. PMID 23598289
- [Derived] Michelsen TM, Tronstad C, Rosseland LA. Blood pressure and cardiac output during caesarean delivery under spinal anaesthesia: a prospective cohort study. BMJ Open. 2021 Jun 14;11(6):e046102. doi: 10.1136/bmjopen-2020-046102. PMID 34127491

RESULTS

PARTICIPANT FLOW:
Groups:
- Carbetocin 100 µg: carbetocin 100 µg : Hemodynamic effect of
- Oxytocin 5 u: oxytocin 5 u : Hemodynamic effect of
- Placebo (NaCl): placebo (NaCl) : Hemodynamic effect of
Period: Overall Study
Arm/Group | Carbetocin 100 µg | Oxytocin 5 u | Placebo (NaCl)
Started | 25 | 26 | 25
Completed | 25 | 26 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbetocin 100 µg | Oxytocin 5 u | Placebo (NaCl) | Total
Number analyzed (Participants) | 25 | 26 | 25 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 26 | 25 | 76
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (3.8) | 35.0 (5.0) | 34.8 (4.0) | 34.5 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 25 | 76
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Norway | 25 | 26 | 25 | 76

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Output
Description: The relative change in CO from baseline at the time of delivery up to 2.5 minutes post delivery.
Time Frame: 2.5 minutes
Measure: Mean (95% Confidence Interval); unit: percentage change in cardiac output
Arm/Group | Carbetocin 100 µg | Oxytocin 5 u | Placebo (NaCl)
Number analyzed (Participants) | 25 | 26 | 25
percentage change in cardiac output | 96 [80 to 111] | 82 [64 to 100] | 43 [35 to 51]

2. Primary Outcome: Arterial Blood Pressure
Description: The mean change in SAP compared with baseline at the time of delivery up to 2.5 minutes post delivery.
Time Frame: 2.5 min
Measure: Mean (95% Confidence Interval); unit: percentage change in arterial blood pres
Arm/Group | Carbetocin 100 µg | Oxytocin 5 u | Placebo (NaCl)
Number analyzed (Participants) | 25 | 26 | 25
percentage change in arterial blood pres | 26 [20 to 31] | 28 [22 to 34] | 16 [9 to 22]

3. Secondary Outcome: Bleeding
Description: The calculated estimated blood loss from delivery until 2 h after intervention
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: ml blood loss
Arm/Group | Carbetocin 100 µg | Oxytocin 5 u | Placebo (NaCl)
Number analyzed (Participants) | 25 | 26 | 25
ml blood loss | 579 (623) | 841 (556) | 853 (518)

ADVERSE EVENTS:
Arm/Group | Carbetocin 100 µg | Oxytocin 5 u | Placebo (NaCl)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 9/25 | 9/26 | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbetocin 100 µg (N=25) | Oxytocin 5 u (N=26) | Placebo (NaCl) (N=25)
Feeling of warmth (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Chest pain (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Nasal congestion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Xerostomia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Metallic taste (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes